CLINICAL TRIAL: NCT01844830
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Parallel-Groups Clinical Trial Comparing The Efficacy And Safety Of Intranasally Administered Kovacaine Mist To Placebo For Anesthetizing Maxillary Teeth In Pediatric Patients
Brief Title: Comparison of Intranasal Kovacaine Mist, and Placebo for Anesthetizing Maxillary Teeth in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR 3-04
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kovacaine Mist (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - Subjects weighing more than 10kg and less than 20kg, will receive 1 spray of 100µL; Subjects weighing more than 20kg and less than 40kg, will receive 2 sprays of 100µL (200µL total); subjects weighting more than 40kg will receive 2 sprays of 200µL (400µL total);
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
- Placebo (Placebo Comparator): Placebo - Subjects weighing more than 10kg and less than 20kg, will receive 1 spray of 100µL; Subjects weighing more than 20kg and less than 40kg, will receive 2 sprays of 100µL (200µL total); subjects weighting more than 40kg will receive 2 sprays of 200µL (400µL total);
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — Intranasally administered regional anesthetic
  Other Names: Kovacaine Mist
  Arms: Kovacaine Mist
Drug: Placebo — Inactive ingredients supplied in identical nasal sprayer
  Other Names: Intranasal administration of inactive ingredients
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of Kovacaine Mist, and Placebo for inducing pulpal anesthesia of the maxillary teeth in pediatric patients.

DETAILED DESCRIPTION:
The study will employ a multi-center, randomized, double-blind, placebo-controlled, parallel-groups design to demonstrate the safety and efficacy of Kovacaine Mist delivered intranasally for inducing pulpal anesthesia of maxillary permanent teeth numbers 4 to 13 (maxillary right second premolar to maxillary left second premolar) or maxillary primary teeth numbers A to J (maxillary right second primary molar to maxillary left second primary molar) sufficient to allow completion of the Study Dental Procedure. The maxillary teeth will be categorized in two subsets, anterior teeth (permanent teeth numbers 6 to 11 and primary teeth numbers C to H) and posterior teeth (permanent teeth numbers 4, 5, 12, 13 and primary teeth numbers A, B, I, J).

The intent is to treat 90 male and female subjects aged 3 to 17 years, inclusive, at 3 study sites, 2:1 randomization within each study site, and an overall goal of 60 subjects treated with Kovacaine Mist and 30 treated with placebo. Subjects will receive Kovacaine Mist or placebo (2:1) according to the kit randomization plan within three dosing strata (100 µL, 200 µL or 400 µL) based on subject weight at entry: subjects weighing 10 to <20 kg, 20 to <40 kg and ≥ 40 kg will be assigned to the 100 µL, 200 µL or 400 µL dose group, respectively. Recruitment will be from diverse pediatric dental patient populations. To ensure adequate representation in the 3 dose/weight groups, each stratum will contain at least 25% of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 3-17 years of age inclusive.
* Need for an operative restorative dental procedure and requiring local anesthesia on a single vital maxillary primary tooth (#A to J) or permanent tooth (#4 to13), with no evidence of pulpal pathology.
* Normal lip, nose, eyelid, and cheek sensation.
* Accompanied and/or represented by a parent or guardian able to comprehend and sign the informed consent document.
* Subject able to understand and provide assent to an age-appropriate subject assent form (as defined by local practice or regulation).
* Patient or parent/guardian able to communicate with the investigator and comply with the requirements of the protocol.
* Patency of the naris on the same side as the tooth undergoing the Study Dental Procedure (the Study Treatment Tooth).

Exclusion Criteria:

* Having received dental care requiring a local anesthetic within the 24 hours preceding study entry.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* History of allergy or hypersensitivity to lidocaine, oxymetazoline, epinephrine, or sulfite preservatives.
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to undergo urine testing on the day of, but prior to, study drug administration to rule out pregnancy.)
* Inadequately controlled thyroid disease of any type.
* Having received any investigational drug (including Kovacaine Mist) and/or participation in any clinical trial within 30 days of study participation.
* Frequent nose bleeds (≥ 5 per month).
* History of congenital or idiopathic methemoglobinemia.
* Presence of an upper respiratory infection and/or fever defined as body temperature ≥100.4° (38°C) on the day of and prior to study drug administration.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Dental Research Loma Linda University School, Loma Linda, California
  - Big Grins, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovacaine Mist | Placebo
Started | 60 | 30
100 µL Dose | 16 | 8
200 µL Dose | 24 | 12
400 µL Dose | 20 | 10
Completed (1 patient in the Kovacaine Mist 200 µL dose group did not finish the study.) | 59 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Mist | Placebo | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (4.2) | 8.1 (3.8) | 8.2 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 32 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 13 | 41
  Not Hispanic or Latino | 32 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 54 | 26 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic.
Description: If the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic and is considered a failure for this outcome.
Time Frame: 100µL dose - at 10 minutes, +3 minute window; for subjects who receive the 200µL or 400µL dose - at 15 minutes, +3 minute window
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Participants | 46 | 16

2. Secondary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic.by Dosage Cohort.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Subjects were in only 1 of 3 dosage cohort. Either 100 µL, 200 µL, or 400 µL.
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Participants
  100 µL: number analyzed (Participants) | 16 | 8
  100 µL | 14 | 7
  200 µL: number analyzed (Participants) | 24 | 12
  200 µL | 14 | 5
  400 µL: number analyzed (Participants) | 20 | 10
  400 µL | 18 | 4

3. Secondary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic. by Age Group (3-5, 6-11, and 12-17 Years Old, Inclusive).
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Patients are grouped by age
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Participants
  3 to 5 years: number analyzed (Participants) | 21 | 10
  3 to 5 years | 17 | 8
  6 to 11 years: number analyzed (Participants) | 23 | 15
  6 to 11 years | 14 | 6
  12 to 17 years: number analyzed (Participants) | 16 | 5
  12 to 17 years | 15 | 2

4. Secondary Outcome: Incidence of Adverse Events (AEs) by Dosage Cohort
Description: Patients with AEs
Time Frame: from baseline to 24 hours following drug administration
Population: Patients grouped by dosage cohort
Measure: Number; unit: Count of participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Count of participants
  100 µL: number analyzed (Participants) | 16 | 8
  100 µL | 12 | 6
  200 µL: number analyzed (Participants) | 24 | 12
  200 µL | 22 | 9
  400 µL: number analyzed (Participants) | 20 | 10
  400 µL | 15 | 7

5. Secondary Outcome: Incidence of Adverse Events (AEs) by Age Group
Description: Patients with AEs
Time Frame: from baseline to 24 hours following drug administration
Population: Patients group by age
Measure: Number; unit: Count of participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Count of participants
  3 to 5 years: number analyzed (Participants) | 21 | 10
  3 to 5 years | 17 | 7
  6 to 11 years: number analyzed (Participants) | 23 | 15
  6 to 11 years | 19 | 11
  12 to 17 years: number analyzed (Participants) | 16 | 5
  12 to 17 years | 13 | 4

6. Secondary Outcome: Results of Naris Examination (NE) - Patency and Ulcerations
Description: The investigators evaluated the treatment naris for patency and ulcerations.
  Patency was evaluated as followed: The nostril not used for dosing study drug was manually occluded and the subject was asked to sniff gently. Airflow in the naris was used to determine if it was patent (yes) or not (no).
  For ulcers, the investigators performed a visual examination for the presence of ulcers and recorded if they were present (yes) or not (no).
Time Frame: 120 minutes post drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
Participants
  Patency (yes) | 59 | 30
  Ulcerations (yes) | 0 | 0

7. Secondary Outcome: Maximum Change From Baseline in Heart Rate
Time Frame: from baseline to 24 hours following drug administration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
bpm | 5.6 (9.09) | 6.9 (9.99)

8. Secondary Outcome: Maximum Change From Baseline in Systolic Blood Pressure
Time Frame: from baseline to 24 hours following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
mmHg | 5.4 (8.78) | 1.0 (8.70)

9. Secondary Outcome: Maximum Change From Baseline in Diastolic Blood Pressure
Time Frame: from baseline to 24 hours following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 60 | 30
mmHg | 8.3 (8.11) | 2.4 (7.09)

10. Secondary Outcome: Results of Naris Examination (NE) - Color
Description: The investigators performed a visual inspection and evaluated the treatment naris for color of the mucosa. The investigator determined what color (Pink, Slightly Red, Red) best matched and recorded the results.
Time Frame: 120 minutes post drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 59 | 30
Participants
  Pink | 52 | 25
  Slightly Red | 6 | 5
  Red | 1 | 0

11. Secondary Outcome: Results of Naris Examination (NE) - Inflammation
Time Frame: 120 minutes post drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 59 | 30
Participants
  No Inflammation | 57 | 29
  Slight Inflammation | 2 | 1
  Inflammation | 0 | 0

12. Secondary Outcome: Results of Naris Examination (NE) - Bleeding
Time Frame: 120 minutes post drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 59 | 30
Participants
  None | 57 | 29
  Slight / Minor | 2 | 1
  Significant / Major | 0 | 0

ADVERSE EVENTS:
Arm/Group | Kovacaine Mist | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30
Other Adverse Events (participants affected / at risk) | 40/60 | 18/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist (N=60) | Placebo (N=30)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 1 — (runny nose)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 6 | 3 — (stinging or burning sensation)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Headache (Nervous system disorders) | 3 | 1
Lacrimation increased (Eye disorders) | 17 | 6 — (tearing or watery eyes)
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Injection Site Pain (General disorders) | 7 | 7
Injection Site Anaesthesia (General disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No